CLINICAL TRIAL: NCT03056222
Title: CardioFocus vs. Contact Force Guided Pulmonary Vein Isolation in Paroxysmal Atrial Fibrillation
Acronym: CF²
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: I-Med-Pro GmbH (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CF2 Rev.1 IMP
Record Dates: First submitted 2017-02-14; First posted 2017-02-17 (Actual); Last update posted 2021-11-19 (Actual); Status verified 2021-11

CONDITIONS: Paroxysmal Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation | interventions — Catheter Ablation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- HeartLight® EGLA (Active Comparator): Participants will be treated with the endoscopically guided laser ablation catheter
  Interventions: Device: Ablation catheter
- Contact Force Sensing Irrigated RF ablation (Active Comparator): Participants will be treated with a contact force sensing irrigated radiofrequency ablation catheter
  Interventions: Device: Ablation catheter

INTERVENTIONS:
Device: Ablation catheter — Ablation of paroxysmal atrial fibrillation

SUMMARY:
The aim of the study is to compare the acute procedure and safety outcomes as well as long term clinical outcomes of 2 groups of patients treated with the HeartLight® Endoscopically Guided Laser Ablation (EGLA) or a commercially available Contact Force Sensing Irrigated Radiofrequency (RF) Ablation Catheter plus, at the operator's discretion, 3D Electroanatomical Mapping (EAM) for the treatment of Paroxysmal Atrial Fibrillation (PAF).

ELIGIBILITY:
Inclusion Criteria:

* Patient must not have undergone a previous ablation for the treatment of PAF
* AF Type - Diagnosed with symptomatic paroxysmal atrial fibrillation (PAF) where PAF is defined as recurrent (two or more) episodes of AF that terminate spontaneously in less than seven days, usually less than 48 hours

Exclusion Criteria:

* Atrial fibrillation secondary to a reversible cause or of non-cardiac origin
* Diagnosed with persistent atrial fibrillation defined as recurrent episodes lasting more than 7 and less than 365 days
* More than 4 electrical cardioversions in the year prior to enrollment but not including cardioversions performed within 48 hours of arrhythmia onset
* Documented left atrial thrombus on imaging
* Cannot be removed from anti-arrhythmic drugs for other reasons than atrial fibrillation
* New York Heart Association (NYHA) functional Class III or Class IV heart failure
* Left ventricular ejection fraction < 30%
* Left atrial size > 55 mm as measured in the parasternal antero-posterior view
* Myocardial infarction within 60 days prior to enrolment
* Woman of childbearing potential who is pregnant, lactating or not using adequate birth control

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 360 (Actual)
Dates: Start 2017-04-10 (Actual); Primary Completion 2021-08-16 (Actual); Study Completion 2021-11-15 (Actual)

PRIMARY OUTCOMES:
Freedom from symptomatic, recurrent atrial fibrillation (AF) off of anti-arrhythmic drugs | 12 months post procedure
  Recurrent AF is defined as any documented episode of AF lasting more than 30 seconds after a blanking period of 90 days post procedure

SECONDARY OUTCOMES:
Acute procedure success | 30 minutes post procedure
  Confirmation of electrical isolation with a circular mapping catheter
Procedure and fluoroscopy time | During procedure
  Time will be taken
Incidence of peri-procedural complications | From procedure to 12 months post procedure
  E.g. major bleeding requiring intervention, phrenic nerve palsy, pericardial tamponade, thrombo-embolic events, pulmonary vein (PV) -stenosis, atrial-to-esophageal fistula, death
Freedom from symptomatic, recurrent Atrial Tachy Arrhythmia (ATA) off of anti-arrhythmic drugs | 12 months post procedure
  Recurrent ATA is defined as any documented episode of ATA lasting more than 30 seconds after a blanking period of 90 days post procedure

CONTACTS AND LOCATIONS:
Overall Officials: Andreas Metzner, PD Dr. med., Principal Investigator — Universitäres Herz- und Gefäßzentrum UKE Hamburg
Locations (11):
- Belgium (2):
  - Hartcentrum OLV Aalst, Aalst
  - Hartcentrum Hasselt Jessa Ziekenhuis, Hasselt
- Nemocnice Na Homolce, Prague, Czechia
- Germany (7):
  - Universitätsklinik Erlangen, Erlangen, Bavaria
  - Isar Herz Zentrum, München, Bavaria
  - St. Vinzenz Hospital Köln, Cologne, North Rhine-Westphalia
  - UKSH, Universitäres Herzzentrum, Lübeck, Schleswig-Holstein
  - Vivantes Klinikum Am Urban, Berlin
  - Asklepios Klinik St. Georg, Hamburg
  - Universitäres Herz- und Gefäßzentrum UKE Hamburg, Hamburg
- Blackpool Victoria Hospital, Blackpool, United Kingdom

IPD SHARING:
Plan to Share IPD: No